CLINICAL TRIAL: NCT03764618
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Study of Fostamatinib Disodium in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia
Brief Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Study of Fostamatinib Disodium in the Treatment of wAIHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-935788-057
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Warm Antibody Autoimmune Hemolytic Anemia
Keywords: wAIHA; Warm Antibody Autoimmune Hemolytic Anemia; Warm Autoimmune Hemolytic Anemia
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fostamatinib (Experimental): Initial dose is 100 mg by mouth (PO) twice a day (bid). At week 4 dose will be increased to fostamatinib 150 mg PO bid if subjects have adequately tolerated the study drug in the opinion of the Investigator.
  Interventions: Drug: Fostamatinib disodium
- Placebo (Placebo Comparator): Initial dose is 100 mg by mouth (PO) twice a day (bid). At week 4 dose will be increased to placebo 150 mg PO bid if subjects have adequately tolerated the study drug in the opinion of the Investigator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib disodium — Fostamatinib (100mg PO bid or 150 mg PO bid)
  The dose may be reduced at any time to a dose as low as fostamatinib 100 mg PO qd or matching placebo if dose limiting adverse events are observed.
  Other Names: R935788; Fostamatinib
  Arms: Fostamatinib
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of fostamatinib in subjects with warm antibody autoimmune hemolytic anemia (wAIHA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a diagnosis of primary or secondary warm Antibody Autoimmune Hemolytic Anemia (wAIHA) as documented by a positive direct antiglobulin test (DAT) specific for anti-IgG or anti-IgA.
2. Have failed or not tolerated at least one prior wAIHA treatment regimen, including steroids, rituximab, azathioprine, cyclophosphamide, cyclosporine, MMF, danazol, vincristine, ESA or splenectomy (folate, iron or other supplements do not fulfill this criterion).
3. Have haptoglobin <LLN or total bilirubin >ULN or lactate dehydrogenase (LDH) >ULN.
4. At screening, subject's hemoglobin level must be ≤9 g/dL OR if hemoglobin value >9 g/dL and <10 g/dL, subject must be on an allowed wAIHA treatment AND the subject must have documented symptoms related to anemia (e.g., weakness, dizziness, fatigue, shortness of breath, chest pain).
5. Karnofsky performance status (KPS) ≥70.
6. Subject's concurrent treatment for wAIHA may consist of no more than two of any of the following agents: azathioprine, steroids, ESAs, mycophenolate mofetil, dapsone or danazol at a stable dose

Exclusion Criteria:

1. Subject with other types of Antibody Autoimmune Hemolytic Anemia (AIHA) (e.g., cold antibody AIHA, cold agglutinin syndrome, mixed type AIHA, or paroxysmal cold hemoglobinuria).
2. Subject has AIHA secondary to autoimmune disease, including systemic lupus erythematosus (SLE), or lymphoid malignancy if the underlying disease is not stable or is not well-controlled on current therapy, per investigator medical judgement.
3. Subject has uncontrolled or poorly controlled hypertension, defined as systolic blood pressure ≥135 mmHg or diastolic blood pressure ≥85 mmHg, whether or not the subject is receiving anti-hypertensive treatment.
4. Subject has one or more of the following laboratory abnormalities at screening: neutrophil count of <1,000/μL or platelet count of <30,000/μL, unless due to Evans syndrome; transaminase levels (i.e., alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) >1.5 x ULN.
5. Has documented active hepatitis B or hepatitis C infection or HIV infection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- United States (26):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Arizona Oncology Associates, PC--HOPE Division, Tucson, Arizona
  - Moores UC San Diego Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Harbor UCLA - Lundquist Institute, Torrance, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Banner MD Anderson Cancer Center at North Colorado Medical Center, Greeley, Colorado
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Affiliated Oncologists, Chicago Ridge, Illinois
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke Cancer Network, Clayton, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Oncology - Baylor Research Institute, Dallas, Texas
  - Clear Lake Specialties, Research Dept., Webster, Texas
  - American Oncology Network Vista Oncology Division, Olympia, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Versiti Wisconsin, Inc., Milwaukee, Wisconsin
  - Marshfield Clinic Cancer Center - Stevens Point, Stevens Point, Wisconsin
- Australia (4):
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital - Cancer Trials Unit, Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (4):
  - Universitätsklinik Innsbruck - Innere Medizin V, Innsbruck
  - Universitätsklinikum Salzburg, 3.Medizin/Onkologie, Salzburg
  - Medizinsche Universität Wien, Vienna
  - Hanusch-Krankenhaus, Vienna
- Belarus (2):
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Belgium (3):
  - Ziekenhuis Network Antwerp, Stuivenberg, Antwerp
  - Universitair Ziekenhuis Antwerpen - Hematologie, Edegem
  - AZ Nikolaas, Sint-Niklaas
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment - Dr Georgi Stranski EAD, Pleven, Clinic of Clinical Haematology, Pleven
  - University Multiprofile Hospital for Active Treatment 'Alexandrovska' EAD, Clinic of Clinical Haematology, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sv. Ivan Rilski' EAD, Clinic of Clinical Hematology, Department of Clinical Hematology, Sofia
  - Specialized Hospital for Active Treatment of Hematological Diseases EAD, Sofia, Clinic of Clinical Haematology, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveta Marina' EAD, Varna, Clinic of Clinical Haematology, Varna
- Canada (3):
  - Hamilton Health Sciences- McMaster University Medical Centre, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Czechia (3):
  - Fakultni nemocnice Brno Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Ostrava Klinika hematoonkologie, Ostrava
  - Ustav Hematologie a Krevni Transfuze, Prague
- Denmark (3):
  - Aalborg University Hopital, Aalborg
  - Aarhus University Hospital - Dept of Hematology, Aarhus N
  - Herlev and Gentofte Hospital, Herlev
- France (7):
  - CHU Angers, Angers
  - Institut d'hématologie de Basse Normandie, CHU Caen, Caen
  - CHU Estaing - Chirurgie digestive et Médecine interne, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - Hôpital Saint Antoine, Paris
  - CHU de Bordeaux - GH Sud- Hôpital Haut Lévêque Service Médecine Interne et Maladies Infectieuses, Pessac
  - CHU Toulouse, IUCT Oncopôle, Toulouse
- Georgia (2):
  - M. Zodelava Hematology Centre, Tbilisi, Tbilisi
  - LTD Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - University of Leipzig Medical Center, Medical Department I - Haematology and Cell Therapy, Medical Oncology, Hemophilia, Leipzig
- Hungary (3):
  - Semmelweis Egyetem, Általános Orvostudományi Kar, I.sz. Belgyógyászati Klinika, Haematológiai Osztály,, Budapest
  - Szabolcs-Szatmár- Bereg Megyei Kórházak és Egyetemi Oktatókórház, Jósa András Oktatókórház, Nyíregyháza
  - Pécsi Tudományegyetem, Klinikai Központ, I.számú Belgyógyászati Klinikai, Hematológiai Tanszék, Pécs
- Italy (5):
  - ASST degli Spedali Civili di Brescia, Ematologia UOC, Brescia
  - Fondazione IRCCS Ca'Granda - Ospedale Maggiore Policlinico di Milano - UO Ematologia, Milan
  - SCDU Ematologia AOU "Maggiore della Carità", Novara
  - Ospedale Maggiore, SC Ematologia - Azienda Sanitaria Universitaria Giuliano Isontina, Trieste
  - ULSS8 Berica Ospedale San Bortolo - Unità Operativa Complessa di Ematologia, Vicenza
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Norway (3):
  - Ålesund Hospital, Ålesund
  - Haukeland University Hospital, Bergen
  - Østfold Hopital, Grålum
- Romania (3):
  - Coltea Clinical Hospital, Bucharest
  - Emergency University Hospital Bucharest, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology Cluj-Napoca, Cluj-Napoca
- Russia (6):
  - State Budgetary Healthcare Institution of Novosibirsk Region "City Clinical Hospital №2", Novosibirsk, Russian Federation
  - National Research Center for Hematology, Moscow
  - Botkin Moscow City Clinical Hospital, Moscow
  - State Budgetary Healthcare Institution of Moscow city "City Clinical Hospital No 40 Department of Healthcare of Moscow city", Moscow
  - State Budgetary Healthcare Institution Oncology Dispensary No. 2 of the Ministry of Health of the Krasnodar Territory, Sochi
  - Regional State Autonomous Healthcare Institution "Tomsk Regional Clinical Hospital", Tomsk
- Serbia (3):
  - University Hospital Medical Center "Bezanijska Kosa", Department of Hematology, Belgrade
  - Clinical Center Nis, Clinic for Hematology, Niš
  - Clinical Centre of Vojvodina, Clinic for Hematology, Novi Sad
- Spain (6):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe - Servicio de Hematología, Valencia
- Ukraine (3):
  - Cherkasy Regional Oncology Dispensary, Hematology Center, Cherkasy
  - City Clinical Hospital № 4, Hematology Center, Dnipro
  - Kyiv City Clinical Hospital №9, hematology department №1, Kyiv
- United Kingdom (5):
  - East Kent Haemophilia Centre, Kent and Canterbury Hospital, Canterbury, Kent
  - Roald Dahl Haemostasis and Thrombosis Centre, Royal Liverpool University Hospital, Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Hammersmith Hospital, London
  - The Royal London Hospital, Bart's Health NHS Trust, London
  - Sandwell and West Birmingham NHS Trust, West Bromwich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fostamatinib: Initial dose is 100 mg by mouth (PO) twice a day (bid). At week 4 dose will be increased to fostamatinib 150 mg PO bid if subjects have adequately tolerated the study drug in the opinion of the Investigator.
  Fostamatinib disodium: Fostamatinib (100mg PO bid or 150 mg PO bid)
  The dose may be reduced at any time to a dose as low as fostamatinib 100 mg PO once a day (qd) or matching placebo if dose limiting adverse events are observed.
Period: Overall Study
Arm/Group | Fostamatinib | Placebo
Started | 45 | 45
Completed | 38 | 34
Not Completed | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fostamatinib | Placebo | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age (years) at Screening
  Years | 56.8 (15.32) | 59.9 (15.70) | 58.4 (15.50)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 29 | 23 | 52
  ≥ 65 years | 16 | 22 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 17 | 18 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 43 | 81
  Black or African American | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Other | 1 | 1 | 2
  Missing | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18
  Czechia | 4 | 2 | 6
  Ukraine | 2 | 2 | 4
  United Kingdom | 0 | 1 | 1
  Belarus | 1 | 1 | 2
  Russia | 5 | 0 | 5
  Spain | 2 | 3 | 5
  Canada | 1 | 1 | 2
  Austria | 2 | 4 | 6
  Netherlands | 0 | 1 | 1
  Belgium | 0 | 1 | 1
  Norway | 1 | 0 | 1
  Italy | 2 | 2 | 4
  Georgia | 2 | 1 | 3
  Australia | 2 | 2 | 4
  Bulgaria | 5 | 10 | 15
  France | 3 | 1 | 4
  Serbia | 1 | 1 | 2
  Germany | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Durable Hemoglobin Response
Description: Proportion of subjects achieving a hemoglobin level ≥ 10 g/dL with an increase from Baseline in hemoglobin level of ≥ 2 g/dL on 3 consecutive available visits during the 24-week treatment period.
Time Frame: 24 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Fostamatinib: Initial dose is 100 mg PO bid. At week 4 dose will be increased to fostamatinib 150 mg PO bid if subjects have adequately tolerated the study drug in the opinion of the Investigator.
  Fostamatinib disodium: Fostamatinib (100mg PO bid or 150 mg PO bid)
  The dose may be reduced at any time to a dose as low as fostamatinib 100 mg PO qd or matching placebo if dose limiting adverse events are observed.
- Placebo: Initial dose is 100 mg PO bid. At week 4 dose will be increased to placebo 150 mg PO bid if subjects have adequately tolerated the study drug in the opinion of the Investigator.
  Placebo: Placebo
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 16 | 12

2. Secondary Outcome: A Hemoglobin Response by Week 24
Description: Proportion of subjects with a hemoglobin response by Week 24.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 21 | 16

3. Secondary Outcome: Change From Baseline in Hemoglobin Level of 2 g/dL or Greater
Description: Proportion of subjects with change from baseline in hemoglobin level of 2 g/dL or greater.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 22 | 16

4. Secondary Outcome: Change in Hemoglobin From Baseline to End of Treatment
Description: Change in mean hemoglobin from baseline to end of treatment.
Time Frame: 24 weeks
Population: Of the 72 completed participants, 11 participants were excluded due to hemoglobin value missing or not being eligible during the evaluation period.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 32 | 29
g/dL | 1.99 (2.095) | 1.99 (2.468)

5. Secondary Outcome: Use of Rescue Antibody Autoimmune Hemolytic Anemia (AIHA) Regimens Use After Week 4
Description: Proportion of subjects free of rescue AIHA regimens used after Week 4.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 18 | 18

6. Secondary Outcome: Change in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F)
Description: Change from Baseline to Week 24 in Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-F). The FACIT-F scale is a short, 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. Each item is rated using a 5-point Likert-type scale. The scale range is 0 to 52, with 0 being the worst possible score and 52 being the best possible score indicating no fatigue. Total Score = [Sum of item scores] x [N of items in subscale] ÷ [N of items answered].
Time Frame: 24 weeks
Population: The analysis population includes the intent-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fostamatinib | Placebo
Number analyzed (Participants) | 39 | 37
score on a scale | 4.1 (12.86) | 2.2 (11.03)

ADVERSE EVENTS:
Time Frame: Up to 30 weeks (-28 days screening, 24 weeks treatment, 2 weeks post treatment follow-up)
Arm/Group | Fostamatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 2/45 | 3/45
Serious Adverse Events (participants affected / at risk) | 15/45 | 17/45
Other Adverse Events (participants affected / at risk) | 42/45 | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib (N=45) | Placebo (N=45)
Warm type hemolytic anemia (Blood and lymphatic system disorders) | 6 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 2
Cold type hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 3
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Hemoglobin decreased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fostamatinib (N=45) | Placebo (N=45)
Warm type hemolytic anemia (Blood and lymphatic system disorders) | 16 | 14
Anemia (Blood and lymphatic system disorders) | 4 | 5
Fatigue (General disorders) | 7 | 5
Asthenia (General disorders) | 4 | 6
Pyrexia (General disorders) | 6 | 3
Oedema peripheral (General disorders) | 3 | 3
Hemoglobin decreased (Investigations) | 8 | 6
Blood pressure increased (Investigations) | 4 | 1
COVID-19 (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Hypertension (Vascular disorders) | 11 | 8
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Jaundice (Hepatobiliary disorders) | 0 | 7
Alanine aminotransferase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Palpitations (Cardiac disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03764618/Prot_SAP_000.pdf